CLINICAL TRIAL: NCT00183508
Title: Developing Group Treatments for Acute Stress Disorder
Brief Title: Behavioral Treatments for Acute Stress Disorder In Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Rose T. Zimering, PhD, Boston Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH064584 (NIH); R21MH064584 (NIH); DATR AD-TS
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Occupational Health; Trauma; Job; CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Cognitive Behavioral Therapy

ARMS (2):
- 1 Cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy
- 2 Psychoeducation (Experimental)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Participants will learn cognitive behavioral strategies for symptom reduction
  Arms: 1 Cognitive behavioral therapy
Behavioral: Psychoeducation — Participants will receive psychoeducation regarding common reactions to traumatic events
  Arms: 2 Psychoeducation

SUMMARY:
This study will develop a treatment for firefighters experiencing symptoms of acute stress disorder (ASD). Effective treatments may reduce immediate symptoms and prevent the development of more chronic conditions, such as post-traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Exposure to traumatic events has reached unprecedented proportions in American society, and the rates of PTSD have risen significantly, particularly among populations with repetitive exposure to critical incidents. The continued threat of attacks against Americans warrants development of preventive interventions to reduce the occurrence of PTSD and its precursor, ASD. This study will determine the effectiveness of a preventive treatment in urban firefighters who have experienced a traumatic event.

Firefighters will undergo an initial assessment that will include an interview and self-report questionnaires to measure depression, anxiety, coping skills, social support, physical health, and work functioning. Following the occurrence of a traumatic work-related event, firefighters will be reassessed. The post-incident assessment will consist of self-report questionnaires that assess ASD symptoms.

Participants who display ASD symptoms will be randomly assigned to one of two groups: the first group will learn cognitive behavioral strategies for symptom reduction, and the second group will receive psychoeducation regarding common reactions to traumatic events. Participants' treatment will last for 12 weeks. Participants will have follow-up assessments 1 and 3 months after the interventional part of the study. Assessments will include clinical scales and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Currently an active duty, nonofficer member of a Boston area fire department
* Willing and able to comply with all study requirements

Exclusion Criteria:

* Pregnancy or plan to become pregnant during the study
* Plan to relocate within 2 months of study entry
* Psychotic symptoms within 30 days prior to study entry
* Experiencing severe depression at study entry OR having suicidal thoughts within 30 days prior to study entry
* Evidence of severe organic impairment that would interfere with participation in the study
* Current alcohol or substance dependence
* Currently awaiting outcome of a court case involving exposure to traumatic events through the fire department

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Primary Completion 2005-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Accute stress disorder symptoms | Measured pre- and post-treatment and at follow-up assessments 1 and 3 months after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rose T. Zimering, PhD, Principal Investigator — Boston Veterans Healthcare System
Locations (1):
- Boston Veterans Healthcare System, Boston, Massachusetts, United States